CLINICAL TRIAL: NCT03907592
Title: Effect of Carnitine Supplementation and Resistance Training on Skeletal Muscle Function in Aging
Brief Title: Effect of Carnitine Supplementation and Resistance Training on Skeletal Muscle Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: Medical University of Gdansk (Other); National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Robert Olek, Associate Professor, Gdansk University of Physical Education and Sport
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DSRiK/10/2017
Record Dates: First submitted 2019-04-06; First posted 2019-04-09 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Sarcopenia
Keywords: L-Carnitine; Resistance training; Magnetic resonance imaging; Muscle function; Aging; Leucine
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L-carnitine Group (Experimental): Group participated in the training protocol and supplemented by 1000 mg L-carnitine-L-tartrate in combination with 3000 mg L-leucine per day throughout 24 weeks.
  Interventions: Dietary Supplement: L-carnitine supplementation; Procedure: Resistance training
- Leucine Group (Experimental): Group participated in the training protocol and supplemented by 4000mg of L-leucine per day throughout 24 weeks.
  Interventions: Dietary Supplement: Leucine supplementation; Procedure: Resistance training
- Control Group (Experimental): Group participated in the training protocol without any supplementation throughout 24 weeks.
  Interventions: Procedure: Resistance training

INTERVENTIONS:
Dietary Supplement: L-carnitine supplementation — Supplementation of 1000 mg L-carnitine-L-tartrate in combination with 3000 mg L-leucine per day throughout the study period.
  Arms: L-carnitine Group
Dietary Supplement: Leucine supplementation — Supplementation of 4000 mg L-leucine per day throughout the study period.
  Arms: Leucine Group
Procedure: Resistance training — Resistance training at the gym, twice a week for 24 weeks (48 training units in total).

SUMMARY:
The primary aim of the current research project is to explore whether nutritional supplementation and resistance training might be combined to produce synergistic effects in the prevention of muscle loss during aging.

A secondary aim of this project is to investigate the effects of carnitine with leucine supplementation, in comparison to carnitine supplementation alone, on muscle strength and body composition.

The hypothesis is that resistance training combined with nutritional supplementation have a more beneficial effect than resistance training alone in the prevention of muscle loss during aging. Leucine stimulates carnitine transport into the muscle cells, which improve mitochondrial capacity. Modification in energetic of skeletal muscle affects the body composition and muscle performance.

DETAILED DESCRIPTION:
The study will be included volunteers - women between 60 - 72 years old (n=60). The patients are randomly assigned to two experimental groups (n=20) and control group (n=20). During the 24-weeks intervention period, Group A undergoes training procedure supplemented with the carnitine and leucine, whilst group B undergoes training procedure supplemented with leucine. At the same time control group go through only training procedure. Measurements are performed before, at the mid-point, and at the end of the intervention period.

Approximately 1 week prior to the experimental trial day, participants perform a familiarization session during which one-repetition maximum (1RM) strength testing is also performed to determine the experimental exercise load. Resistance exercise training is performed twice weekly on non-consecutive days (Monday+Thursday, or Tuesday+Friday) for 24-weeks under direct supervision by a research assistant. Prior to a training session subjects are required to perform warm - up on the treadmill (walk) and static stretching, after each session - cool down on the cycle ergometer and static stretching. Resistance exercise for each session consisted of 6 exercises: horizontal seated leg press, seated chest press, leg extension, shoulder press, lat pull-down seated row, seated cable row First two weeks of training consist of 3 sets of 10-12 repetitions and are keeping exercises at 65% of 1 repetition maximum (1RM). After this period training consists of 3 sets of 6-8 repetitions and is progressing to 80% of 1RM. The 1RM is re-evaluated every 2 weeks, and the training load is adjusted accordingly. The exercise program follows the recommended guidelines for older adults by the American College of Sports Medicine and the National Strength and Conditioning Association.

ELIGIBILITY:
Inclusion Criteria:

* aged-matched, no chronic disease, doctor's note about the lack of restrictions to perform resistance exercises

Exclusion Criteria:

* diabetes, liver, heart and renal diseases, gastric problems, as well as using the vitamin supplements

Ages: 60 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
Volumetric changes in knee extensor muscle | Values at baseline will be compared to values recorded at 12 and at 24 weeks after supplementation and training procedure.
  Volumetric examination of cross section area (CSA) of knee extensor muscles determined by a 1.5 T MRI scanner.

SECONDARY OUTCOMES:
Changes in the strength of muscle knee extensor | Values at baseline will be compared to values recorded at 12 and at 24 weeks after supplementation and training procedure.
  Maximal isometric knee extensor peak torques determined by the dynamometer (Biodex System 4 Pro).
Changes in Lean Body Mass | Values at baseline will be compared to values recorded at 12 and at 24 weeks after supplementation and training procedure.
  Lean Body Mass measured by dual-energy X-ray absorptiometry (DXA).

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Olek, PhD, Principal Investigator — Gdansk University of Physical Education and Sport
Locations (1):
- University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland